CLINICAL TRIAL: NCT02446574
Title: Phase I /II Study of Postoperative Chemoradiation in Patients With Node-positive Esophageal Squamous Cell Carcinoma
Brief Title: Postoperative Chemoradiation in Patients With Node-positive Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zefen Xiao, Clinical Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-27/230
Record Dates: First submitted 2015-04-26; First posted 2015-05-18 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Esophageal Neoplasms
Keywords: chemoradiation; dose escalation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A (Experimental): During the Phase I it will administered weekly paclitaxel(dose escalation) and cisplatin with concurrent radiation therapy
  During the Phase II it will administered weekly paclitaxel(dose according to phase I) and cisplatin with concurrent radiation therapy
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Paclitaxel — starting dose 20mg/m2 qw
  Other Names: taxel
Drug: Cisplatin — dose 25mg/m2 qw
  Other Names: platimum
Radiation: Radiation — 60Gy/2Gy/30f

SUMMARY:
This is a unicentered phase I/II study to explore the dose of paclitaxel and cisplatin with radiation therapy, and to document the adverse events for further clinical trial.

DETAILED DESCRIPTION:
Although preoperative chemoradiation therapy followed by surgery is the most common approach for patients with resectable esophageal cancer, the considerable number of esophageal cancer patients received operation as the first treatment modality. Accordingly, postoperative treatments have been playing an important role because of the poor survival rates of the patients with pathologically positive lymph nodes who have been treated with resection alone. The investigators have proved the value of prophylactic radiation therapy after radical esophagectomy for esophageal carcinoma with positive lymph node metastases under the conventional 2-dimensional radiotherapy methods in subset analysis of prospective randomized clinical trial. For patients with positive lymph nodes, 5 year survival after surgery alone was 28.4%, median overall survival was 24 months, recurrence occurred 34.6% in mediastinal lymph nodes，13.3% in supraclavicular lymph nodes，10% in abdominal lymph nodes. Distant metastases occurred in 21% patients. Adjuvant radiotherapy significantly reduced the recurrence in mediastinal lymph nodes(13.4%), supraclavicular lymph nodes (6.1%). However distant metastases rate increased to 30.7%. Chemotherapy may be vital for these patients. Chen reported that the 5 year overall survival rates for the chemoradiotherapy group and radiotherapy group were 47.4% and 38.6% (P=0.03). Based on the investigators' studies, treatment failure occurred in 8% patients because of celiac metastases. Small radiation field by omitting celiac axis lymph node basin may ensure 5-6 cycles of concurrent chemotherapy for lower toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. KPS≥70
2. Diagnosis of pathologically positive lymph node thoracic esophageal cancer
3. Complete resection
4. Adequate organ function:

Hematopoietic Absolute granulocyte count at least 1,500/mm^3 Platelet count at least 150,000/mm^3 Hemoglobin at least 10 g/dL Hepatic Not specified Renal Creatinine no greater than 1.5 mg/dL AND/OR Creatinine clearance at least 65 mL/min Calcium no greater than 11 mg/dL Cardiovascular No uncontrolled heart disease No uncontrolled hypertension

Exclusion Criteria:

1. Uncontrolled diabetes
2. Interval between surgery and adjuvant therapy more than 3 months
3. Sign of recurrence on CT scan or ultrasound or PET-CT No palpable supraclavicular lymph nodes or involvement after cytology needle aspiration No lymph nodes greater than 1 cm on CT scan
4. With Weight loss greater than 10% from baseline
5. With other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
6. Be pregnant

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of weekly paclitaxel and cisplatin with concurrent radiation(Phase I endpoint) | 3 months

SECONDARY OUTCOMES:
Toxicities according to the Common Terminology Criteria for Adverse Events version 3.0. | 18 months
Overall Survival survival of weekly paclitaxel and cisplatin with concurrent radiation(Phase II endpoint) | 60 months
Disease-free survival of weekly paclitaxel and cisplatin with concurrent radiation(Phase II endpoint) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Zefen Xiao, Professor, Principal Investigator — Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Science
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Rizk N, Venkatraman E, Park B, Flores R, Bains MS, Rusch V; American Joint Committee on Cancer staging system. The prognostic importance of the number of involved lymph nodes in esophageal cancer: implications for revisions of the American Joint Committee on Cancer staging system. J Thorac Cardiovasc Surg. 2006 Dec;132(6):1374-81. doi: 10.1016/j.jtcvs.2006.07.039. PMID 17140960
- [Result] Korst RJ, Rusch VW, Venkatraman E, Bains MS, Burt ME, Downey RJ, Ginsberg RJ. Proposed revision of the staging classification for esophageal cancer. J Thorac Cardiovasc Surg. 1998 Mar;115(3):660-69; discussion 669-70. doi: 10.1016/S0022-5223(98)70332-0. PMID 9535455
- [Result] Rice TW, Blackstone EH, Rybicki LA, Adelstein DJ, Murthy SC, DeCamp MM, Goldblum JR. Refining esophageal cancer staging. J Thorac Cardiovasc Surg. 2003 May;125(5):1103-13. doi: 10.1067/mtc.2003.170. PMID 12771884
- [Result] Hagen JA, DeMeester SR, Peters JH, Chandrasoma P, DeMeester TR. Curative resection for esophageal adenocarcinoma: analysis of 100 en bloc esophagectomies. Ann Surg. 2001 Oct;234(4):520-30; discussion 530-1. doi: 10.1097/00000658-200110000-00011. PMID 11573045
- [Result] Igaki H, Kato H, Tachimori Y, Nakanishi Y. Prognostic evaluation of patients with clinical T1 and T2 squamous cell carcinomas of the thoracic esophagus after 3-field lymph node dissection. Surgery. 2003 Apr;133(4):368-74. doi: 10.1067/msy.2003.76. PMID 12717353
- [Result] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Result] Rice TW, Adelstein DJ, Chidel MA, Rybicki LA, DeCamp MM, Murthy SC, Blackstone EH. Benefit of postoperative adjuvant chemoradiotherapy in locoregionally advanced esophageal carcinoma. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1590-6. doi: 10.1016/s0022-5223(03)01025-0. PMID 14666038
- [Result] Liu HC, Hung SK, Huang CJ, Chen CC, Chen MJ, Chang CC, Tai CJ, Tzen CY, Lu LH, Chen YJ. Esophagectomy for locally advanced esophageal cancer, followed by chemoradiotherapy and adjuvant chemotherapy. World J Gastroenterol. 2005 Sep 14;11(34):5367-72. doi: 10.3748/wjg.v11.i34.5367. PMID 16149148
- [Result] Hsu PK, Huang CS, Wang BY, Wu YC, Hsu WH. Survival benefits of postoperative chemoradiation for lymph node-positive esophageal squamous cell carcinoma. Ann Thorac Surg. 2014 May;97(5):1734-41. doi: 10.1016/j.athoracsur.2013.12.041. Epub 2014 Mar 6. PMID 24612702
- [Result] Chen J, Pan J, Liu J, Li J, Zhu K, Zheng X, Chen M, Chen M, Liao Z. Postoperative radiation therapy with or without concurrent chemotherapy for node-positive thoracic esophageal squamous cell carcinoma. Int J Radiat Oncol Biol Phys. 2013 Jul 15;86(4):671-7. doi: 10.1016/j.ijrobp.2013.03.026. PMID 23773390
- [Result] Xiao ZF, Yang ZY, Liang J, Miao YJ, Wang M, Yin WB, Gu XZ, Zhang DC, Zhang RG, Wang LJ. Value of radiotherapy after radical surgery for esophageal carcinoma: a report of 495 patients. Ann Thorac Surg. 2003 Feb;75(2):331-6. doi: 10.1016/s0003-4975(02)04401-6. PMID 12607634